CLINICAL TRIAL: NCT05259540
Title: Effect of Compound Kushen Injection Combined With Pabolizumab in the Treatment of Cervical Adenocarcinoma: A Phase II Single-arm Clinical Study
Brief Title: Effect of Compound Kushen Injection Combined With Pabolizumab in the Treatment of Cervical Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210164
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer
Keywords: PD1; PD-L1; Cervical adenocarcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- compound kushen injection combined with pabolizumab (Experimental): compound kushen injection 20ml/day and pabolizumab 200mg/21 days
  Interventions: Drug: compound kushen injection combined with pabolizumab

INTERVENTIONS:
Drug: compound kushen injection combined with pabolizumab — compound kushen injection 20ml/day and pabolizumab 200mg/21 days, both drugs are given intravenously
  Other Names: experience group

SUMMARY:
In the past few decades, the incidence of endocervical adenocarcinomas (ECAs) has been on the rise both in absolute numbers and overall proportion in cervical cancers. ECAs remain a significant public health problem despite advances in treatment options. Patients with ECA have a poorer survival rate than patients with squamous cell carcinoma (SCC), especially in patients with metastatic tumors. In the newly published 2020 World Health Organization (WHO) Classification of Female Genital Tumors, ECAs are subclassified into human papillomavirus-associated (HPVA) and human papillomavirus-independent (HPVI) groups. Meanwhile, PD-1/PD-L1 immunotherapy has been approved for the treatment of advanced cervical cancer, but there are still many deficiencies. Therefore, the investigators plan to use the new classification of female genital tumors and conduct a clinical trial to explore the safety and effectiveness of compound kushen injection combined with pabolizumab in the treatment of metastatic, recurrent, persistent cervical adenocarcinoma.

DETAILED DESCRIPTION:
In this study, PD-1 inhibitors (pabolizumab) combined with compound kushen injection were used to treat metastatic, recurrent, persistent cervical adenocarcinoma, and the efficacy and safety of the two drugs were evaluated.

Participants who meet the requirements will sign the informed consent and be enrolled voluntarily. This project is a single-arm study without a control group. Forty-two patients are expected to be enrolled.

Two scoring systems, the combined positive score (CPS) and the tumor proportion score (TPS), are used for evaluation of PD-L1 expression of solid tumors. Through the measurable changes in the size of the lesions, the investigators can understand the changes of the disease. The primary endpoints were PFS and ORR. Whenever, for whatever reason, the subject does not complete the clinical trial observation, is considered to be an abscission case. When the subject falls off, the investigators must fill in the reason for the fall off in the CRF, and contact the subject as much as possible, complete the items that can be evaluated, and record the time of the last medication to prepare for the analysis of its efficacy and safety. The CRF should be kept for future reference.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥ 18 yrs and ≤75 yrs;
2. Patients volunteered to participate in this study, signed informed consent, good compliance, and cooperated with follow-up;
3. The subjects' damage caused by other treatments has been recovered (NCI CTCAE version 5.0 grade ≤ grade 1), ECOG score ≤ 2 points;
4. Expected survival is longer than 3 months;
5. Pathological diagnosis of cervical advanced adenocarcinoma (PD-L1 positive, TPS score ≥1%; CPS score ≥1);
6. Evaluable lesions: CT scan of tumor lesions ≥5mm in length, CT scan of lymph node lesions ≥10mm in length, and scan layer thickness not greater than 5mm (refer to RECIST 1.1);
7. The first diagnosis was confirmed by pathology and / or cytology to be metastatic, or recurrent, persistent cervical adenocarcinoma (mainly refers to tumors remaining or progressing at least 3 months after initial radiotherapy or concurrent chemoradiotherapy), and the patient can no longer accept Surgery or chemoradiation;
8. Subject agrees to take blood sample;
9. Subjects can provide formalin-fixed, paraffin-embedded tumor tissue samples for subsequent related testing (optional);
10. A.Complete blood count: hemoglobin (Hb) ≥90g/L ; absolute neutrophil count (ANC) ≥1.0×109/L ; platelets >=100×109/L B. Biochemical test standards: a. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 times the upper limit of normal value (ULN). If with liver metastases, ALT and AST ≤ 5 × ULN; b. Total bilirubin (TBIL) ≤ 1.5 × ULN; c. Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 60ml / min; d. Doppler ultrasound evaluation: left ventricular ejection Blood fraction (LVEF) ≥ the lower limit of normal value (50%).
11. Women of childbearing age should agree that contraception (such as an intrauterine device, contraceptive, or condom) must be used during the study and within 3 months after the last dose; a serum or urine pregnancy test must be negative within 14 days of study enrollment and must be Non-lactating patients. Sign written informed consent before conducting any research-related procedures.

Exclusion Criteria:

1. People who are known to be allergic to compound kushen injection and pabolizumab or to active or inactive ingredients of drugs with similar chemical structures to compound kushen injection and pabolizumab.
2. Symptomatic, uncontrolled brain metastases or pia meningeal metastases.
3. No imaging scan is required to confirm brain-free metastases; patients with spinal cord compression may still be considered if they have received targeted treatment and have evidence of clinical stability of the disease for at least> 28 days (controlled central nervous system metastasis must be in the study Have received treatment such as radiation or chemotherapy for at least 1 month; patients must not have new symptoms related to central nervous system lesions or symptoms that indicate disease progression, and patients either take a stable dose of hormones or do not need to take hormones).
4. Underwent major surgery within 3 weeks before the study began, or any surgical effects that have not recovered after surgery, or received chemotherapy.
5. Received> 20% bone marrow palliative radiotherapy 1 week before enrollment.
6. Have aggressive cancers other than cervical cancer (except fully treated basal or squamous cell skin cancer within 2 years before enrollment).
7. Patient has a previous or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
8. Suffering from a serious or uncontrolled illness, including but not limited to:

1. Uncontrollable nausea and vomiting, inability to swallow research drugs, and any gastrointestinal disorders that may interfere with the metabolism of the drug.

2. Active viral infections such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.

3. Uncontrolled major seizures, unstable spinal cord compression, superior vena cava syndrome, or other mental illnesses that prevent patients from signing informed consent.

4. Immunodeficiency (except splenectomy), or other diseases that the investigator believes may expose patients to high-risk toxicity.

9. History of bleeding and thrombosis:

1. Any CTCAE Grade 2 bleeding event within 3 months prior to screening, or CTCAE Grade 3 and above bleeding events within 6 months prior to screening.
2. History of gastrointestinal bleeding or clear gastrointestinal bleeding tendency within 6 months before screening. Such as: esophageal varices at risk of bleeding, focal lesions of locally active ulcers, or fecal occult blood +.
3. Have active bleeding or coagulopathy, have a tendency to bleed, or are receiving thrombolytic or anticoagulant therapy.
4. Patients need anticoagulation with drugs such as warfarin or heparin.
5. Patients need long-term antiplatelet therapy (eg aspirin, clopidogrel).
6. Thrombosis or embolism events in the past 6 months, such as: cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism.

10. Serious cardiovascular history:

1. NYHA (New York Heart Association) Grade 3 and 4 congestive heart failure.
2. Suffering from unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening.
3. Arrhythmias requiring therapeutic intervention (patients taking beta-blockers or digoxin can be enrolled).
4. CTCAE≥ grade 2 valvular heart disease.

11. Poorly controlled hypertension (systolic blood pressure> 150 mmHg or diastolic blood pressure> 100 mmHg).

12. Other laboratory inspection abnormalities:

1. Hyponatremia (sodium <130 mmol / L); baseline serum potassium <3.5 mmol / L (before entering the study, potassium supplements can be used to restore serum potassium above this level).
2. Abnormal thyroid function, and drugs cannot maintain thyroid function within normal range.

13. Any previous or current disease, treatment, or laboratory abnormality that may interfere with the results of the study, affect the patient's full participation in the study, or the investigator believes that the patient is not suitable to participate in the study; the patient may not receive platelets within 4 weeks before the study drug begins Red blood cell infusion.

14. Patients who are pregnant or breastfeeding, or plan to become pregnant during study treatment.

15. Corrected QTc interval (QTc)> 450 milliseconds; if the patient has a prolonged QTc interval, but the investigator evaluates that the reason for the prolongation is a pacemaker (and no other cardiac abnormalities), it is necessary to discuss with the investigator to determine whether the patient is suitable Group study.

16. With any active autoimmune disease or have a history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo or asthma has been completely relieved in childhood and do not need any intervention after adulthood could be included; Asthma patient who need bronchodilators for medical intervention cannot be included) 17. Treatment with other immunosuppressive medications, systemic or topical corticosteroids (>10 mg daily prednisone or equivalent) within 14 days before enrollment.

18. With a history of severe allergic reaction to other monoclonal antibodies. 19. Evidence of central nervous system metastasis (such as brain edema requiring hormone intervention, or brain metastasis progression). Patients who have previously received treatment for brain or meningeal metastasis and persistently stable (MRI) for at least 1 month thus stopped systemic hormone therapy (dose > 10mg/ prednisone or other therapeutic hormones) for more than 2 weeks can be included.

20. Have previously received any PD-1/PD-L1 inhibitor treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 weeks
  To evaluate the objective response rate (CR + PR) of compound kushen injection combined with pabolizumab in patients with cervical adenocarcinoma.

SECONDARY OUTCOMES:
PFS | 6 months
  progression-free survival
DCR | 6 months
  disease control rate
DOR | 6 months
  duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Lili Chen, MD, Principal Investigator — Zhejiang University School of Medicine Women's Hospital
Locations (1):
- Lili Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen L, Niu Y, Wan X, Yu L, Zhang X, Strickland AL, Dong L, Zhou F, Lu W. Clinicopathological features and outcomes in gastric-type of HPV-independent endocervical adenocarcinomas. BMC Cancer. 2021 Oct 11;21(1):1095. doi: 10.1186/s12885-021-08792-7. PMID 34635081
- [Background] Chen L, Lucas E, Zhang X, Liu Q, Zhuang Y, Lin W, Chen H, Zhou F. Programmed death-ligand 1 expression in human papillomavirus-independent cervical adenocarcinoma and its prognostic significance. Histopathology. 2022 Jan;80(2):338-347. doi: 10.1111/his.14552. Epub 2021 Oct 13. PMID 34455625
- [Background] Frenel JS, Le Tourneau C, O'Neil B, Ott PA, Piha-Paul SA, Gomez-Roca C, van Brummelen EMJ, Rugo HS, Thomas S, Saraf S, Rangwala R, Varga A. Safety and Efficacy of Pembrolizumab in Advanced, Programmed Death Ligand 1-Positive Cervical Cancer: Results From the Phase Ib KEYNOTE-028 Trial. J Clin Oncol. 2017 Dec 20;35(36):4035-4041. doi: 10.1200/JCO.2017.74.5471. Epub 2017 Nov 2. PMID 29095678
- [Background] Chung HC, Ros W, Delord JP, Perets R, Italiano A, Shapira-Frommer R, Manzuk L, Piha-Paul SA, Xu L, Zeigenfuss S, Pruitt SK, Leary A. Efficacy and Safety of Pembrolizumab in Previously Treated Advanced Cervical Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2019 Jun 10;37(17):1470-1478. doi: 10.1200/JCO.18.01265. Epub 2019 Apr 3. PMID 30943124